CLINICAL TRIAL: NCT06683521
Title: Immunologic Basis of Food Protein-Induced Enterocolitis Syndrome
Acronym: INFINITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-01346; U01AI170836-01 (NIH)
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Food Protein-Induced Enterocolitis Syndrome
Keywords: Allergy; FPIES; Food protein-induced enterocolitis syndrome; Food; Diagnosis
MeSH Terms: conditions — Hypersensitivity; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will be sequentially enrolled into 3 cohorts of 24 each.
  The first cohort will undergo Low Dose OFC to 300 mg food protein. Following interim analysis of Low Dose OFC outcomes in cohort 1, the Low Dose OFC serving size may be amended or continued at 300 mg food protein for cohort 2 & 3 based on pre-specified criteria.
  Interventions: Other: Supervised Low-Dose Oral Food Challenge (OFC); Other: At-Home Low-Dose Oral Food Challenge (OFC); Other: Supervised High-Dose Oral Food Challenge (OFC)
- Cohort 2 (Experimental): Participants will be sequentially enrolled into 3 cohorts of 24 each.
  Following interim analysis of Low Dose OFC outcomes in cohort 1, Low-Dose OFC may be continued at 300 mg food protein or be amended for cohort 2 and 3 based on pre-specified criteria.
  Interventions: Other: Supervised Low-Dose Oral Food Challenge (OFC); Other: At-Home Low-Dose Oral Food Challenge (OFC); Other: Supervised High-Dose Oral Food Challenge (OFC)
- Cohort 3 (Experimental): Participants will be sequentially enrolled into 3 cohorts of 24 each.
  Following interim analysis of Low Dose OFC outcomes in cohort 1, Low-Dose OFC may be continued at 300 mg food protein or be amended for cohort 2 and 3 based on pre-specified criteria.
  Interventions: Other: Supervised Low-Dose Oral Food Challenge (OFC); Other: At-Home Low-Dose Oral Food Challenge (OFC); Other: Supervised High-Dose Oral Food Challenge (OFC)

INTERVENTIONS:
Other: Supervised Low-Dose Oral Food Challenge (OFC) — All participants will undergo a supervised Low Dose OFC (300 mg food protein or amended) on Day 1.
Other: At-Home Low-Dose Oral Food Challenge (OFC) — Participants who tolerate the Day 1 Low Dose OFC will undergo a daily Low-Dose OFC (300 mg food protein or amended) at home on Days 2-7.
Other: Supervised High-Dose Oral Food Challenge (OFC) — Participants who tolerate the Days 1-7 Low Dose OFC will undergo a supervised High Dose OFC (maximum 3000 mg food protein) on Day 8.

SUMMARY:
This is a phase I multicenter clinical trial that aims to find the optimal dose for conducting a novel low-dose, multi-day oral food challenge (OFC) protocol for diagnosing food protein-induced enterocolitis syndrome (FPIES). Individuals ages 1-60 years with a history of suspected or confirmed FPIES will be eligible for enrollment. Recruitment is expected to occur over 3 years.

DETAILED DESCRIPTION:
At the time of enrollment, participants will undergo screening (Visit 0) and complete a baseline gastrointestinal symptom diary.

At Visit 1 (Day 1), participants will undergo a supervised Low Dose OFC to their FPIES trigger. Those who react will be considered low-threshold reactors and recommended to continue strict avoidance of their FPIES trigger.

For participants who do not react at the Day 1 Low Dose OFC, continued participation involves a daily home challenge on Days 2-7. Participants will be provided with a diary to monitor symptoms. If objective or persistent subjective symptoms develop, participants will be advised to contact the study team before consuming any further doses.

Participants will return for Visit 2 on Day 8. Those who reported symptoms that led to discontinuation of the home challenge will undergo biospecimen collection. Those who tolerated the Day 1 supervised and Days 2-7 home challenges will undergo a High Dose OFC to their suspected FPIES trigger. Those who tolerate this challenge will be considered to have outgrown their FPIES and instructed to introduce the food regularly at home. Those who react will be considered high-threshold reactors and advised to continue strict avoidance of their FPIES trigger and continue routine allergy care.

ELIGIBILITY:
Inclusion Criteria:

* Provision of appropriate consent and/or assent
* Age 1-60 years
* Suspected or confirmed FPIES diagnosis
* Reported convincing FPIES reaction (per criteria in 2017 FPIES guidelines) within: (Children <18 years of age: The past 6-36 months) (Adults age >18 years: The past 6 months-10 years)
* Individuals of childbearing potential practicing sexual abstinence or using effective methods of contraception during study participation
* English-speaking

Exclusion Criteria:

* Past severe FPIES defined as hospitalization due to an acute FPIES reaction with neurological compromise or requiring life support
* Acute FPIES reaction in the past 6 months
* Frequent gastrointestinal symptoms: nausea, abdominal pain, reflux, heartburn, emesis, diarrhea, constipation per participant or guardian report or as evidenced by FPIES Symptoms Score (FPIES-SS)
* Current active eosinophilic gastrointestinal disorders, inflammatory bowel disease, gastroesophageal reflux disease, or any other chronic gastrointestinal condition
* Poorly controlled atopic dermatitis at screening per PI discretion
* Poorly controlled or severe asthma/wheezing at screening, defined by at least one of the following criteria: 1: History of two or more systemic corticosteroid courses within six months of screening or one course of systemic corticosteroids within three months of screening to treat asthma/wheezing; 2: Prior intubation/mechanical ventilation for asthma/wheezing; 3: One hospitalization or ED visit for asthma/wheezing within six months of screening; and 4: Inhaled corticosteroid (ICS) dosing of >500 mcg daily fluticasone (or equivalent ICS based on National Heart, Lung, and Blood Institute (NHLBI) dosing chart).
* IgE-mediated food allergies where the trigger has not been identified
* Inability to discontinue prohibited medications for 7 days prior to the screening visit and lasting for the duration of study participation unless indicated for use as rescue medication
* Personal or family history of prolonged QT syndrome
* Personal history of arrhythmia
* Current diagnosis of arterial hypertension
* Current diagnosis of cardiovascular disease
* Current diagnosis of any chronic autoimmune disease
* Current diagnosis of liver disease
* Primary or secondary immunodeficiency
* Phenylketonuria (PKU) (ondansetron tablets may contain phenylalanine)
* Use of systemic steroids within 30 days of screening
* Chemotherapy, radiotherapy, or any systemic immunosuppressive drugs in the past 12 months
* Use of biologic drugs or allergen-specific immunotherapy by any route in the past 12 months
* Inability to defer routine immunizations or passive immunization with immune globulin for the duration of participation in the study
* Allergy to any of the following medications: ondansetron (Zofran), dolasetron (Azemet), granisetron (Kytril), or palonosetron (Aloxi)
* Pregnancy or breastfeeding
* Current or past medical problems or findings from the physical examination or screening evaluation not listed above, which, in the opinion of the investigator(s), may pose additional risks from study participation, interfere with the participant's ability to comply with study requirements, and/or impact the quality or interpretation of the data obtained from the study

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of individuals with active FPIES who develop FPIES symptoms during the optimal Low Dose multi-day OFC (Days 1-7) | Up to Day 7

SECONDARY OUTCOMES:
Percentage of participants who meet criteria for intravenous fluid (IVF) resuscitation among those who develop FPIES symptoms during Low Dose multi-day OFC (Days 1-7)[Time Frame: Up to Day 7] | Up to Day 7
Percentage of participants treated with oral ondansetron among those who develop FPIES symptoms during Low Dose multi-day OFC | Up to Day 7
Percentage of participants treated with parenteral ondansetron among those who develop FPIES symptoms during Low Dose multi-day OFC | Up to Day 7
Percentage of participants with hypotension among those who develop FPIES symptoms during Low Dose multi-day OFC (Days 1-7) | Up to Day 7
  Hypotension defined as: a systolic blood pressure (mmHg): age 1-10: Systolic <70+(age in years x 2); 11 years or older: <90 mmHg.
Percentage of participants with reactions treated in the Emergency Department (ED) among those who develop FPIES symptoms during Low Dose multi-day OFC (Days 1-7) | Up to Day 7
Number of participants with reactions resulting in overnight admission to ED/Hospital among those who develop FPIES symptoms during Low Dose multi-day OFC (Days 1-7) | Up to Day 7
Median number of emesis episodes among those who develop FPIES symptoms during Low Dose multi-day OFC (Days 1-7) | Up to Day 7
Median maximum severity of abdominal pain score (assessed with the FPIES-SS) among those who develop FPIES symptoms during Low Dose multi-day OFC (Days 1-7) | Up to Day 7
  The FPIES-SS is a 15-item questionnaire assessing gastrointestinal symptoms. Each item is rated on a scale from 0-10. The scores corresponding to responses to each question are averaged over the number of days the symptoms were recorded; the final score is calculated by adding averages and dividing by 15 (the number of scorable items). The final score ranges from 0-10; higher scores indicate greater severity of gastrointestinal symptoms.
Median time to discharge during Day 1 Supervised Low Dose OFC among those who develop FPIES symptoms during Low Dose multi-day OFC | Day 1
  Measure taken on Day 1.
Median time to resolution of symptoms during Day 1 Supervised Low Dose OFC among those who develop FPIES symptoms during Low Dose multi-day OFC | Day 1
  Measure taken on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nowak-Wegrzyn, MD, PhD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Jaffe Food Allergy Institute at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
At time of publication, the study team will share primary data (flow cytometry and sequence data) through the National Institute of Allergy and Infectious Diseases (NIAID)-supported repository: "ImmPort." Datasets will be made available immediately after the primary manuscripts from the research have been accepted for publication, with no end date. Upon reasonable request, the investigator who proposed to use the data will be able to access via ImmPort. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: No end date.
Access Criteria: Upon reasonable request, the investigator who proposed to use the data will be able to access via ImmPort.